CLINICAL TRIAL: NCT02701699
Title: A Feasibility Study of Hypoxia Imaging in Patients With Lung Cancer Using Positron Emission Tomography (PET) With 18F-Fluoroazomycin Arabinoside (18F-FAZA)
Brief Title: 18F-Fluoroazomycin Arabinoside (18F-FAZA) in Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 13-6528-C
Record Dates: First submitted 2014-12-09; First posted 2016-03-08 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; FAZA PET Imaging; Lung Radiotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18-F-FAZA Scan (Experimental): All patients enrolled in this study will receive a FAZA PET Scan prior to their first radiation therapy fraction
  Interventions: Biological: 18-F-FAZA

INTERVENTIONS:
Biological: 18-F-FAZA — All patients enrolled in this study will receive a FAZA PET Scan prior to their first radiation therapy fraction

SUMMARY:
The purpose of this study is to look for low levels of oxygen (hypoxia) in lung cancer using a positron emission tomography (PET) scan. Hypoxia can influence how lung cancer grows and responds to treatments like radiotherapy and chemotherapy. The use of PET scans to measure hypoxia may be better and simpler than the approaches used previously. This study will assess whether or not PET scans can provide useful information about hypoxia in lung cancer.

In this study, a radiotracer called Fluoroazomycin Arabinoside (FAZA) will be used to measure hypoxia in the patient's tumour. FAZA has already been used in many cancers including lung cancer. Patients who consent to participate in this trial will receive 1 FAZA PET Scan prior to their first radiotherapy treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with stage II or III lung cancer (both NSCLC and SCLC) qualifying for radiotherapy to the primary tumor, with or without treatment of mediastinal or hilar lymph nodes
3. Intention to treat using radiotherapy according to the current treatment policies of the PMH Lung Group
4. Concurrent systemic therapy allowed
5. A negative serum pregnancy test within the two week interval immediately prior to PET-CT imaging, in women of child-bearing age
6. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

1. Previous radiotherapy to intended treatment volumes.
2. Previous systemic therapy
3. Active malignancy other than lung cancer
4. Unable to remain supine for more than 60 minutes
5. Pregnancy
6. Age less than 18 years old
7. Failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with lung cancer using the PET tracer FAZA to image primary tumor hypoxia prior to treatment with radiotherapy | 5 years
Number of patients with lung cancer using 4D (gated) and static PET imaging of FAZA uptake | 5 years

SECONDARY OUTCOMES:
Proportion of the volume of injected FAZA tracer taken up in the tumor prior to treatment with radiotherapy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Sun, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada